CLINICAL TRIAL: NCT03148678
Title: Scrutinizing and Promoting Mindfulness Via New Technologies: Smartphone-based Assessment and Micro-intervention and Functional Magnetic Resonance Imaging (fMRI) (-Neurofeedback)
Brief Title: Scrutinizing and Promoting Mindfulness Via New Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Korea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: GRNP_2013S1A2A2035364_1_2
Record Dates: First submitted 2017-03-24; First posted 2017-05-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Mindfulness; Stress; Mood; Working Memory
Keywords: Emotional reactivity; Cognitive flexibility
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: A combination of sequential (mindfulness vs. mind wandering intervention) and parallel design (contingent vs. non-contingent RT-fMRI-NF)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness first; Contingent RT-fMRI-NF (Experimental): Participants start with the mindfulness intervention followed by the mind wandering intervention. The arm type "experimental" refers to contingent RT-fMRI-NF, during which participants are provided with contingent RT-fMRI-NF of their own brain activity.
  Interventions: Behavioral: Mindfulness; Other: Contingent RT-fMRI-NF; Behavioral: Mind Wandering
- Mindfulness first; Non-Contingent Neurofeedback (Sham Comparator): Participants start with the mindfulness intervention followed by the mind wandering intervention. The arm type "sham comparator" refers to non-contingent RT-fMRI-NF, during which participants are provided with sham RT-fMRI-NF of brain activity of previously recorded subject.
  Interventions: Behavioral: Mindfulness; Other: Sham RT-fMRI-NF; Behavioral: Mind Wandering
- Mind wandering first; Contingent Neurofeedback (Experimental): Participants start with the mind wandering intervention followed by the mindfulness intervention. The arm type "experimental" refers to contingent RT-fMRI-NF, during which participants are provided with contingent RT-fMRI-NF of their own brain activity.
  Interventions: Behavioral: Mindfulness; Other: Contingent RT-fMRI-NF; Behavioral: Mind Wandering
- Mind wandering first; Non-Contingent Neurofeedback (Sham Comparator): Participants start with the mind wandering intervention followed by the mindfulness intervention. The arm type "sham comparator" refers to non-contingent RT-fMRI-NF, during which participants are provided with sham RT-fMRI-NF of brain activity of previously recorded subject.
  Interventions: Behavioral: Mindfulness; Other: Sham RT-fMRI-NF; Behavioral: Mind Wandering

INTERVENTIONS:
Behavioral: Mindfulness — Subjects are provided with smartphone-based mindfulness intervention.
Other: Contingent RT-fMRI-NF — Subjects are provided with contingent RT-fMRI-NF of their own brain activity.
  Arms: Mind wandering first; Contingent Neurofeedback; Mindfulness first; Contingent RT-fMRI-NF
Other: Sham RT-fMRI-NF — Subjects are provided with sham RT-fMRI-NF of brain activity of previously recorded subject.
  Arms: Mind wandering first; Non-Contingent Neurofeedback; Mindfulness first; Non-Contingent Neurofeedback
Behavioral: Mind Wandering — Subjects are provided with smartphone-based mind wandering intervention.

SUMMARY:
The overall goal of the outlined study is to scrutinize and to promote mindfulness via new technologies using a combination of smartphone-based assessment and micro-interventions, fMRI and real-time fMRI-neurofeedback.

DETAILED DESCRIPTION:
The overall goal of the outlined study is to scrutinize and to promote mindfulness via new technologies using a combination of smartphone-based assessment and micro-interventions, fMRI and real-time fMRI-neurofeedback. More specifically, we aim to i) evaluate whether smartphone-based micro-interventions affect mindfulness, stress, and mood, ii) evaluate whether mindfulness, its neural substrate, and related mental and physiological functions can be modified by training volitional control over brain activity by means of real-time functional magnetic resonance imaging neurofeedback (RT-fMRI-NF), iii) differentiate neural activation patterns during mindfulness vs. mind wandering.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness
* Ability to participate in study procedures

Exclusion Criteria:

* Color-Blindness
* Present or past psychological or psychiatric therapy
* Presence of cardiovascular disease
* History of major cerebral injury
* Medical MRI contraindication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) Signal assessed by MRI | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Blood oxygenation level dependent (BOLD) signal assessed via functional magnetic resonance imaging
State mindfulness assessed by State Mindfulness Scale | Daily, during smartphone-based micro-interventions (duration: 10 days); on 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last smartphone-based micro-intervention days)
  State mindfulness, assessed via State Mindfulness Scale (SMS)
Subjective stress reactivity assessed by Visual Analog Scale | Daily, during smartphone-based micro-interventions (duration: 10 days); on 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last smartphone-based micro-intervention days)
  Subjective stress reactivity, assessed via Visual Analog Scale (VAS)
Subjective mood assessed by Multidimensional Mood State Questionnaire | Daily, during smartphone-based micro-interventions (duration: 10 days); on 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last smartphone-based micro-intervention days)
  Subjective mood, assessed via Multidimensional Mood State Questionnaire (MDMQ)

SECONDARY OUTCOMES:
Emotional reactivity assessed by emotion recognition task | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via emotion recognition task
Working Memory assessed by N-back task test | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via N-back task (visual single-3-back with letters as stimuli)
Cognitive flexibility assessed by computer version of Wisconsin card sorting Task test | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via computer version of Wisconsin card sorting task (WCST)

OTHER OUTCOMES:
Respiration Signal assessed by sensor | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via sensor
Trait mindfulness assessed by Mindful Attention Awareness Scale | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via Mindful Attention Awareness Scale (MAAS)
Heart rate assessed by sensor | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via sensor
Subjective stress reactivity assessed by Perceived Stress Scale test | On 1 day, which is the laboratory assessment day (scheduled 1 day subsequent to the last of the 10 smartphone-based micro-intervention days)
  Assessed via Perceived Stress Scale (PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Hwan Lee, Ph.D., Principal Investigator — Korea University
Locations (2):
- Korea University, Seoul, South Korea
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HC, Lee JH. Spectral dynamic causal modeling of mindfulness, mind-wandering, and resting-state in the triple network using fMRI. Neuroreport. 2022 Mar 23;33(5):221-226. doi: 10.1097/WNR.0000000000001772. PMID 35287148